CLINICAL TRIAL: NCT03485209
Title: Open Label Phase 2 Study of Tisotumab Vedotin for Locally Advanced or Metastatic Disease in Solid Tumors
Brief Title: Efficacy and Safety Study of Tisotumab Vedotin for Patients With Solid Tumors
Acronym: innovaTV 207
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Genmab (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNTV-001; C5721001; innovaTV 207 (Other: Alias Study Number); 2023-503812-34-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2018-03-08; First posted 2018-04-02 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Exocrine Pancreatic Cancer; Carcinoma, Squamous Cell of Head and Neck
Keywords: Colorectal cancer; NSCLC; sqNSCLC; CRC; Pancreatic cancer; Head and neck cancer; Seattle Genetics; HNSCC
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Pancreatic Neoplasms; Head and Neck Neoplasms | interventions — tisotumab vedotin; pembrolizumab; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: Tisotumab Vedotin - Q3W Schedule (Experimental): Tisotumab Vedotin on Day 1 of every 21-day cycle in participants with various solid tumors in 2L+
  Interventions: Drug: tisotumab vedotin
- Part B: Tisotumab Vedotin - 3Q4W Schedule (Experimental): Tisotumab Vedotin on Days 1, 8, and 15 of 28-day cycle in participants with various solid tumors in 2L+
  Interventions: Drug: tisotumab vedotin
- Part C: Tisotumab Vedotin - 2Q4W Schedule (Experimental): Tisotumab Vedotin on Days 1 and 15 of every 28-day cycle in participants with HNSCC or sqNSCLC in 2L+
  Interventions: Drug: tisotumab vedotin
- Part D: Tisotumab Vedotin Combination Therapy - Q3W Schedule (Experimental): Tisotumab Vedotin + pembrolizumab + (carboplatin or cisplatin). Given on Day 1 of every 21-day cycle in participants with various solid tumors in 1L HNSCC or sqNSCLC
  Interventions: Drug: tisotumab vedotin; Drug: pembrolizumab; Drug: carboplatin; Drug: cisplatin
- Part E: Tisotumab Vedotin - 2Q4W Schedule (Experimental): Tisotumab Vedotin on Days 1 and 15 of every 28-day cycle in participants with HNSCC in the second- or third-line setting
  Interventions: Drug: tisotumab vedotin
- Part F: Tisotumab Vedotin Combination Therapy - Q2W Schedule (Experimental): Tisotumab Vedotin + pembrolizumab. Tisotumab Vedotin given on Days 1, 15, and 29 of every 6-week cycle. Pembrolizumab given on Day 1 of every 6-week cycle in participants with HNSCC in the first line setting
  Interventions: Drug: tisotumab vedotin; Drug: pembrolizumab
- Part G: Tisotumab Vedotin Combination Therapy - Q2W Schedule (Experimental): Tisotumab Vedotin + pembrolizumab + carboplatin. Tisotumab Vedotin and carboplatin given on Days 1, 15, and 29 of every 6-week cycle. Pembrolizumab given on Day 1 of every 6-week cycle in participants with HNSCC in the first line setting
  Interventions: Drug: tisotumab vedotin; Drug: pembrolizumab; Drug: carboplatin

INTERVENTIONS:
Drug: tisotumab vedotin — Given into the vein (IV; intravenously)
  Other Names: TIVDAK
Drug: pembrolizumab — 200mg or 400mg given by IV
  Other Names: KEYTRUDA®
  Arms: Part D: Tisotumab Vedotin Combination Therapy - Q3W Schedule; Part F: Tisotumab Vedotin Combination Therapy - Q2W Schedule; Part G: Tisotumab Vedotin Combination Therapy - Q2W Schedule
Drug: carboplatin — AUC 5mg/mL per minute or AUC 3.3mg/mL per minute given by IV
  Arms: Part D: Tisotumab Vedotin Combination Therapy - Q3W Schedule; Part G: Tisotumab Vedotin Combination Therapy - Q2W Schedule
Drug: cisplatin — 100mg/m^2 given by IV
  Arms: Part D: Tisotumab Vedotin Combination Therapy - Q3W Schedule

SUMMARY:
This trial will study tisotumab vedotin to find out whether it is an effective treatment alone or with other anticancer drugs for certain solid tumors and what side effects (unwanted effects) may occur. There are seven parts to this study.

* In Part A, participants will receive tisotumab vedotin every 3 weeks (3-week cycles).
* In Part B, participants will receive tisotumab vedotin on Days 1, 8, and 15 every 4-week cycle.
* In Part C, participants will receive tisotumab vedotin on Days 1 and 15 of every 4-week cycle.
* In Part D, participants will be given treatment on Day 1 of every 3-week cycle.
* Participants in Part D will get tisotumab vedotin with either:

  * Pembrolizumab or,
  * Pembrolizumab and carboplatin, or
  * Pembrolizumab and cisplatin
* In Part E, participants will receive tisotumab vedotin on Days 1 and 15 of every 4-week cycle.
* In Part F, participants will receive tisotumab vedotin on Days 1, 15, and 29 of every 6-week cycle. Participants in Part F will get tisotumab vedotin with pembrolizumab.
* In Part G, participants will receive tisotumab vedotin on Days 1, 15, and 29 of every 6-week cycle. Participants in Part G will get tisotumab vedotin with pembrolizumab and carboplatin.

The objectives of the study have been achieved. Therefore, the study will transition to a long-term extension phase (LTEP).

* In LTEP, participants still receiving clinical benefit based on the investigator's assessment and remaining on treatment may continue receiving treatment.
* Participants will still receive tisotumab vedotin with either:

  * Pembrolizumab or,
  * Pembrolizumab and carboplatin, or
  * Pembrolizumab and cisplatin

DETAILED DESCRIPTION:
The primary goal of this trial is to assess the activity, safety, and tolerability of tisotumab vedotin for the treatment of selected solid tumors. Patients will be treated with single agent tisotumab vedotin or tisotumab vedotin in combination with other anticancer agents. Patients who meet eligibility criteria will be enrolled into cohorts based on tumor type. Tumor types to be evaluated include colorectal cancer, squamous non-small cell lung cancer (sqNSCLC), exocrine pancreatic adenocarcinoma, and head and neck squamous cell carcinoma (HNSCC).

ELIGIBILITY:
Inclusion Criteria:

* Parts A, B, and C

  * Relapsed, locally-advanced or metastatic colorectal or pancreatic cancer, sqNSCLC, or HNSCC participants who are not candidates for standard therapy.
  * All participants must have experienced disease progression on or after their most recent systemic therapy.
  * Colorectal cancer (closed to enrollment): participants must have received prior therapy with each of following agents, if eligible: a fluoropyrimidine, oxaliplatin, irinotecan, and/or bevacizumab. Participants should have received no more than 3 systemic regimens in the metastatic setting.
  * sqNSCLC (closed to enrollment): Participants with NSCLC must have predominant squamous histology. Participants must have received prior therapy with a platinum-based treatment and a checkpoint inhibitor (CPI), if eligible. Participants should have received no more than 3 lines of systemic therapy in the metastatic setting.

    * Participants eligible for a tyrosine kinase inhibitor should have received such therapy. These participants should have received no more than 4 lines of systemic therapy in the metastatic setting.
  * Exocrine pancreatic adenocarcinoma (closed to enrollment): Participants with exocrine pancreatic adenocarcinoma must have predominant adenocarcinoma histology. Participants must have received prior therapy with a gemcitabine-based or 5FU-based regimen, if eligible, and should have received no more than 1 systemic regimen in the unresectable or metastatic setting.
  * HNSCC (closed to enrollment): Participants with HNSCC in Part C must have received prior therapy with a platinum-based regimen and/or a checkpoint inhibitor (CPI), if eligible, and must have experienced disease progression following such therapy. Participants should have received no more than 3 systemic lines of therapy in the recurrent or metastatic setting.
* Part E

  * Part E is closed to enrollment.
  * Participants with HNSCC must have experienced disease progression on or after their most recent systemic therapy. Participants should have received no more than 1 or 2 systemic lines of therapy in the recurrent/metastatic setting as specified below. Participants must have received a platinum-based regimen and a PD-(L)1 inhibitor.
* Parts D, F, and G

  * Part D and F are closed to enrollment. Part G will enroll only participants with HNSCC.
  * Participants with HNSCC must have received no previous systemic therapy in the recurrent or metastatic disease setting.
  * Part D only

    * Participants with NSCLC must have histologically or cytologically documented squamous cell NSCLC and must have received no previous systemic therapy for metastatic disease or radiation therapy to the lung that is > 30 Gy within 6 months of the first dose of study treatment.
    * PD-L1 biomarker expression as determined by a PD-L1 IHC assay should be available
  * Part F only

    * Participants must have CPS ≥1 by local PD-L1 IHC assay to be eligible for enrollment. Participants must be able to submit a tissue sample for retrospective PD-L1 testing. Tissue may be fresh biopsy or archival, collected within 2 years of Cycle 1 Day 1.
  * Part G only

    * Part G cohort was not opened.
    * Non-EU eligibility criteria: No CPS requirement for the cohort evaluating tisotumab vedotin in combination with pembrolizumab and carboplatin.
    * EU-specific eligibility criteria: Participants must have a CPS ≥1 by local PD-L1 IHC assay.
    * Participants must be able to submit a tissue sample for retrospective PD-L1 testing. Tissue may be fresh biopsy or archival, collected within 2 years of Cycle 1 Day 1.
* Baseline measurable disease as measured by RECIST v1. 1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.

Exclusion Criteria:

* Participants with primary neuroendocrine or sarcomatoid histologies. For HNSCC, participants may not have a primary site of nasopharynx or salivary gland.
* Active bleeding conditions
* Clinically significant cardiac disease including stable angina, acute myocardial infraction 6 months prior to screening
* Ocular surface disease at the time of enrollment (Note: cataract is not considered active ocular surface disease for this protocol)
* Other cancer: known past or current malignancy other than inclusion diagnosis.
* Uncontrolled tumor-related pain
* Inflammatory lung disease. Participants with pulmonary disease are allowed if systemic steroids and long-term oxygen are not required
* Peripheral neuropathy greater than or equal to Grade 2
* Active brain metastasis
* Ongoing clinically significant toxicity associated with prior treatment (including radiotherapy or surgery).
* Part D, F, and G Only: Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) (Parts A, B, C, D, E, F, and G) | Up to approximately 3 years
  Proportion of patients who achieve a confirmed complete response (CR) or partial response (PR) according to RECIST v1.1 as assessed by the investigator

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to approximately 3 years
  Type, severity, and relatedness of adverse events. An AE is any untoward medical occurrence in a subject or clinical investigational subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Confirmed and Unconfirmed ORR | Up to approximately 3 years
  Proportion of patients who achieve a CR or PR according to RECIST v1.1 as assessed by the investigator
Disease Control Rate (DCR) | Up to approximately 3 years
  Proportion of patients who achieve a confirmed CR or PR according to RECIST v1.1 as assessed by the investigator, or meet the stable disease (SD) criteria at least once after start of study treatment at a minimum interval of 12 weeks
Duration of Response (DOR) | Up to approximately 3 years
  Time from the first documentation of objective response to the first documentation of PD or death due to any cause, whichever comes first, as assessed by the investigator
Time to Response (TTR) | Up to approximately 1 year
  Time from the start of study treatment to the first documentation of objective response, as assessed by investigator
Progression-free survival (PFS) | Up to approximately 3 years
  Time from the start of study treatment to the first documentation of PD according to RECIST v1.1 or death due to any cause, whichever comes first, as assessed by the investigator
Overall Survival (OS) | Up to approximately 4 years
  Time from the start of study treatment to date of death due to any cause
Cmax | Through 30-37 days following the last dose; up to approximately 3 years
  Maximum observed plasma concentration
Ctrough | Through 30-37 days following the last dose; up to approximately 3 years
  Observed plasma concentration at the end of the dosing interval
Incidence of anti-therapeutic antibodies (ATAs) | Through 30-37 days following the last dose; up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (167):
- United States (118):
  - UCSD Medical Center - Encinitas, Encinitas, California
  - UC San Diego Medical Center - La Jolla (Jacobs Medical Center / Thornton Pavilion), La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCSD Koman Family Outpatient Pavilion, La Jolla, California
  - UC San Diego/Moores Cancer Center, La Jolla, California
  - UCSD Shiley Eye Institute, La Jolla, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center- Hillcrest, San Diego, California
  - UC San Diego Health - Rancho Bernardo, San Diego, California
  - Stanford Cancer Center South Bay, San Jose, California
  - UCSD Medical Center - Vista, Vista, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Eye Center of Northern Colorado, Fort Collins, Colorado
  - Cancer Care & Hematology - Fort Collins, Fort Collins, Colorado
  - Cancer Care & Hematology - Greeley, Greeley, Colorado
  - Cancer Care & Hematology - Loveland, Loveland, Colorado
  - Simlow Cancer Hospitalat Yale-New Haven, New Haven, Connecticut
  - Yale-New Haven Hospital- Yale Cancer Center, New Haven, Connecticut
  - C/O Thomas Ferenez.RPh,BCOP,Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Family Focus Eye Care - Gainesville, Gainesville, Florida
  - UF Health Davis Cancer Pavilion and Shands Med Plaza, Gainesville, Florida
  - UF Health Shands Cancer Hospital, Gainesville, Florida
  - UF Health Shands Hospital, Gainesville, Florida
  - Family Focus Eye Care - Lake City, Lake City, Florida
  - Moffitt Cancer Center McKinley Hospital, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Richard M Schulze Family Foundation Outpatient Center at McKinley Campus, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Investigational Drug Service, Emory University Clinic, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - UChicago Medicine - River East, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Kishwaukee Hospital, DeKalb, Illinois
  - Primary Healthcare Associates, Flossmoor, Illinois
  - UChicago Medicine at Ingalls - Flossmoor, Flossmoor, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Delnor Hospital, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Primary Healthcare Associates, Harvey, Illinois
  - UChicago Medicine Ingalls Memorial, Harvey, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - The University of Chicago Medicine Center for Advanced Care Orland Park, Orland Park, Illinois
  - Primary Healthcare Associates, Tinley Park, Illinois
  - UChicago Medicine at Ingalls - Tinley Park, Tinley Park, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Community Health Network, Inc., Indianapolis, Indiana
  - The University of Kansas Cancer Center ,Investigational Drug Services, Fairway, Kansas
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute Pharmacy, Louisville, Kentucky
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - The Eye Care Institute, Louisville, Kentucky
  - Norton Audubon Hospital, Louisville, Kentucky
  - Norton Cancer Institute, Audubon Hospital Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Norton Cancer Institute, Brownsboro Hospital Campus, Louisville, Kentucky
  - John Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts Eye and Ear Infirmary(MEEI), Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ophthalmic Consultants of Boston Inc (OCB), Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Oncology Research, HealthPartners Institute, Saint Louis Park, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University - Investigational Drug Service Pharmacy, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - MSK Basking Ridge., Basking Ridge, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack., Commack, New York
  - MSK Westchester., Harrison, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care (74th Street)., New York, New York
  - MSK Nassau., Uniondale, New York
  - North Carolina Basnight Cancer Hospital Infusion Pharmacy, Chapel Hill, North Carolina
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - Investigational Chemotherapy Service, Durham, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Atrium Health Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Atrium Health Wake forest Baptist, Winston-Salem, North Carolina
  - OHSU Knight Cancer Institute, Beaverton, Beaverton, Oregon
  - OHSU Knight Cancer Institute, Gresham, Gresham, Oregon
  - OHSU Knight Cancer Institute, Northwest Portland, Portland, Oregon
  - OHSU Knight Cancer Institute, East Portland, Portland, Oregon
  - OHSU Center for Health and Healing 2, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - Oregon Health and Science University Research Pharmacy Services, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - OHSU Knight Cancer Institute, Tualatin, Tualatin, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Renovatio Clinical., The Woodlands, Texas
  - Cancer Center IDS Pharmacy, Charlottesville, Virginia
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
  - UVA Health System; Attention: GI Team, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Cross Cancer Institute, Edmonton, Alberta, Canada
- France (15):
  - CHRU de Besançon- Hopital Jean Minjoz, Besançon, Doubs
  - Laboratoire Oriade Noviale Medipole, Bourgoin
  - Laboratoire Oriade Noviale Tixier, Bourgoin
  - The Centre Léon Bérard, Lyon
  - Lbmms Du Chu de Lyon, Lyon
  - CEPCM/CHU Timone, Batiment 3 -1er etage, Marseille
  - Hopital prive du Confluent S.A.S., Nantes
  - L'hôpital Privé du Confluent - Pharmacie, Nantes
  - Synlab Bourgogne Pont de Vaux, Pont-de-Vaux
  - Laboratoire Cerballiance Portes Les Valence, Portes-lès-Valence
  - Hôpital Foch Pharmacie - Essais Cliniques, Suresnes
  - Hôpital Foch, Suresnes
  - LBM UNIBIO Jean Herve Lebras, Tain-l'Hermitage
  - Laboratoire Trevoux-Dyomedea Neolab, Trévoux
  - Gustave Roussy, Villejuif
- Germany (3):
  - Vincentius-Diakonissen-Klinken Gag Augenklinik, Karlsruhe
  - Vincentius-Diakonissen-Kliniken gAG Medizinische Klinik 2, Karlsruhe
  - Vincentius-Diakonissen-Klinken Gag Radiologisches Institut, Karlsruhe
- Italy (14):
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori Dino Amadori- IRST S.r.l, Meldola (Fc), Emilia-Romagna
  - Oncologia Medica, Ospedale Civile S. Maria delle Croci, Ravenna, Emilia-Romagna
  - IRST IRCCS - Farmacia Oncologica, Meldola (FC), Forli-cesena
  - UOC Oncologia Medica, Rome, Lazio
  - U.O. Oncologia, Brescia, Lombardy
  - Istituto Europeo di Oncologia, Milan, MI
  - Ospedale Cervesi di Cattolica-AUSL Romagna, Cattolica, RN
  - Ospedale degli Infermi -AUSL Romagna, Rimini, RN
  - PO Ospedale degli Infermi Faenza, AUSL Romagna, Faenza
  - Ospedale Umberto I di Lugo, AUSL della Romagna, SSR Emilia-Romagna, Lugo
  - AOU Università degli studi della Campania Luigi Vanvitelli, Policlinico di Napoli, Napoli
  - Azienda Ospedaliera Universitaria - Universita della Campania Luigi Vanvitelli, Napoli
  - Ospedale S.Jacopo di Pistoia, AUSL Toscana centro, SST, Pistoia
  - Farmacia Oncologica c/o Ospedale S.Maria delle Croci-AUSL Romagna, Ravenna
- Spain (9):
  - Institut Catala D 'Oncologia-Hospital Germans Trias I Pujol,Servicio de Oncologia Medica, Barcelona, Badalona
  - ALTHAIA, Xarxa Assistencial Universitaria de Manresa., Manresa, Barcelona
  - Hospital Quironsalud Barcelona Instituto Oncologico Baselga, Barcelona, Catalonia
  - Hospital Quiron Salud Barcelona Plaza, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitario Dexeus - Grupo Quirónsalud, Barcelona
  - Fundació Hospital Universitari Vall d'Hebron - Institut de Recerca, Barcelona
  - Institut Catala d'Oncologia (ICO BADALONA), Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
- United Kingdom (7):
  - Clinical Research Facility - Clinical Research Facility, London, London, CITY of
  - Guy's and St Thomas' NHS Foundation Trust - Guy's Hospital, London, London, CITY of
  - Guys and St Thomas Hospital, London, Other
  - Pharmacy Stores (CCR5916) - The Royal Marsden, Sutton, Surrey
  - The Royal Marsden NHS Foundation Trust (RM)., London
  - Royal Marsden Hospital NHS Foundation Trust - HNTU, Sutton
  - The Royal Marsden NHS Foundation trust (RM), Sutton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Feng S, Gunawan R, Passey C, Voellinger J, Polhamus D, Gerritsen A, O'Day C, Carret AS, Soumaoro I, Gupta M, Hanley WD. Exposure-safety Markov modeling of ocular adverse events in patient populations treated with tisotumab vedotin. J Pharmacokinet Pharmacodyn. 2025 Oct 3;52(5):55. doi: 10.1007/s10928-025-10003-w. PMID 41044356
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNTV-001